CLINICAL TRIAL: NCT06168357
Title: Role of Abbreviated MRI in Follow-up of Hepatocellular Carcinoma Following Locoregional Treatment.
Brief Title: Role of Abbreviated MRI in Follow-up of Hepatocellular Carcinoma .
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Nour Mokhles Farah, Assistant Lecturer, Assiut University
Other Study IDs: Role of MRI in HCC
Record Dates: First submitted 2023-12-05; First posted 2023-12-13 (Actual); Last update posted 2023-12-13 (Actual); Status verified 2023-11

CONDITIONS: Hepatocellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

SUMMARY:
Role of ADC value and DWI in abbreviated MRI compared to post-contrast CT in follow-up of HCC after TACE.

DETAILED DESCRIPTION:
Hepatocellular carcinoma (HCC) is the 5th most common cancer in the world and the most common in Egypt .

Trans-arterial chemoembolization (TACE) is the treatment recommended for unresectable HCC according to Barcelona clinic liver cancer staging and is widely used .

HCC is nourished only by the hepatic artery, so TACE causes ischemia and coagulative necrosis. However; viable neoplastic tissue residual may be seen after TACE. Assessment of post-TACE tumor response is important in determining treatment success and in guiding future therapy .

Many studies have assessed the diagnostic performance of multiphasic contrast-enhanced computed tomography (CT) and magnetic resonance imaging (MRI) in diagnosis of HCC with noted higher sensitivity of MRI compared to CT. CT or MRI are recommended for assessment of response after treatment as well .

Diffusion-weighted imaging (DWI) and apparent diffusion coefficient (ADC) are functional MRI techniques that detect signal changes in tissues due to water proton motion. The intact membranes of viable tumor cells restrict water diffusion, whereas necrotic tumor cells with disrupted cell membranes exhibit increased water diffusion and which differentiate the biological activity of HCC

ELIGIBILITY:
Inclusion Criteria:

* Patients who underwent TACE for unresectable HCC with patent portal vein based on Doppler, no ascites, and satisfactory liver function.

Age between 20-year old and 85-year old

Exclusion Criteria:

* Estimated GFR less than 60 Previous history of severe allergic reaction to the iodinated contrast agent Patients with claustrophobia who can't undergo MR examination. Patients having cochlear implants or cardiac pacemaker

Ages: 20 Years to 85 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients who underwent TACE for unresectable HCC with patent portal vein based on Doppler, no ascites, and satisfactory liver function.
  Age between 20-year old and 85-year old.
Sampling Method: Non-Probability Sample
Enrollment: 55 (Estimated)
Dates: Start 2024-01 (Estimated); Primary Completion 2025-09-30 (Estimated); Study Completion 2027-09-30 (Estimated)

PRIMARY OUTCOMES:
Correlation between tumor enhancement in arterial phase expressed as Hounsfield unit number and ADC value. | Baseline
  correlation between tumor enhancement in arterial phase expressed as Hounsfield unit number and ADC value.

REFERENCES:
- [Result] Liu Z, Fan JM, He C, Li ZF, Xu YS, Li Z, Liu HF, Lei JQ. Utility of diffusion weighted imaging with the quantitative apparent diffusion coefficient in diagnosing residual or recurrent hepatocellular carcinoma after transarterial chemoembolization: a meta-analysis. Cancer Imaging. 2020 Jan 6;20(1):3. doi: 10.1186/s40644-019-0282-9. PMID 31907050
- [Result] European Association for the Study of the Liver. EASL Clinical Practice Guidelines: Management of hepatocellular carcinoma. J Hepatol. 2018 Jul;69(1):182-236. doi: 10.1016/j.jhep.2018.03.019. Epub 2018 Apr 5. No abstract available. Erratum In: J Hepatol. 2019 Apr;70(4):817. doi: 10.1016/j.jhep.2019.01.020. PMID 29628281
- [Result] Sung PS, Choi MH, Yang H, Lee SK, Chun HJ, Jang JW, Choi JY, Yoon SK, Choi JI, Lee YJ, Bae SH. Diffusion-Weighted Magnetic Resonance Imaging in Hepatocellular Carcinoma as a Predictor of a Response to Cisplatin-Based Hepatic Arterial Infusion Chemotherapy. Front Oncol. 2020 Nov 19;10:600233. doi: 10.3389/fonc.2020.600233. eCollection 2020. PMID 33330098
- [Result] Gluskin JS, Chegai F, Monti S, Squillaci E, Mannelli L. Hepatocellular Carcinoma and Diffusion-Weighted MRI: Detection and Evaluation of Treatment Response. J Cancer. 2016 Jul 13;7(11):1565-70. doi: 10.7150/jca.14582. eCollection 2016. PMID 27471573
- [Result] Wang WT, Yang L, Yang ZX, Hu XX, Ding Y, Yan X, Fu CX, Grimm R, Zeng MS, Rao SX. Assessment of Microvascular Invasion of Hepatocellular Carcinoma with Diffusion Kurtosis Imaging. Radiology. 2018 Feb;286(2):571-580. doi: 10.1148/radiol.2017170515. Epub 2017 Sep 22. PMID 28937853
- [Result] Ludwig JM, Camacho JC, Kokabi N, Xing M, Kim HS. The Role of Diffusion-Weighted Imaging (DWI) in Locoregional Therapy Outcome Prediction and Response Assessment for Hepatocellular Carcinoma (HCC): The New Era of Functional Imaging Biomarkers. Diagnostics (Basel). 2015 Nov 30;5(4):546-63. doi: 10.3390/diagnostics5040546. PMID 26854170
- [Result] Surov A, Pech M, Omari J, Fischbach F, Damm R, Fischbach K, Powerski M, Relja B, Wienke A. Diffusion-Weighted Imaging Reflects Tumor Grading and Microvascular Invasion in Hepatocellular Carcinoma. Liver Cancer. 2021 Feb;10(1):10-24. doi: 10.1159/000511384. Epub 2021 Jan 27. PMID 33708636